CLINICAL TRIAL: NCT05912751
Title: Acute Responses of Postural Alignment, Kinematic Synergy, and Intermuscular Coherence to Postural Muscle Facilitation (Retrospective)
Acronym: PPMvsRCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radford University (Other)
Responsible Party: Principal Investigator, Stephen Glass, Assistant Professor, Radford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-288-RUC (Retrospective)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Posture; Musculoskeletal Equilibrium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Then Foam Roll (Other): This arm (sequence) will first complete the exercise intervention promoting muscular engagement resisting gravitational collapsing tendencies, then the control intervention involving self-myofascial release of muscle groups not thought to resist gravitational collapse.
  Interventions: Other: Exercise Then Foam Roll
- Foam Roll Then Exercise (Other): This arm (sequence) will first complete the control intervention involving self-myofascial release of muscle groups not thought to resist gravitational collapse, then the exercise intervention promoting muscular engagement resisting gravitational collapsing tendencies.
  Interventions: Other: Foam Roll Then Exercise

INTERVENTIONS:
Other: Exercise Then Foam Roll — Participants in AB will perform the experimental (exercise) intervention first and the control (foam rolling) intervention second.
  Other Names: AB
  Arms: Exercise Then Foam Roll
Other: Foam Roll Then Exercise — Participants in BA will perform the control (foam rolling) intervention first and the experimental (exercise) intervention second.
  Other Names: BA
  Arms: Foam Roll Then Exercise

SUMMARY:
Postural alignment is often intervened upon in health, fitness, and physical medicine settings. Despite a long tradition in this area, current notions of optimal or normal posture are superficial and often logically inconsistent. A recent attempt to reconcile diverging opinions about good posture proposes that alignment be considered in relation to individual joints' natural tendencies to collapse under gravity. This theory allows different maladaptive postures to be described in terms of functional deficits and compensatory adaptations at the muscular level. Working within this type of theory, postural interventions may be able to account for comparative advantages in maintaining alignment between different muscle systems. This would represent a step forward from current practices, which usually attempt to force arbitrary alignment patterns indiscriminately.

The current study presents motion capture and electromyography (EMG) data evaluating the effects of two interventions on individual participants' bipedal standing alignment patterns with respect to the gravitational collapsing tendencies referenced above. Additional outcomes included functional grouping of muscle activation signals (via intermuscular coherence) and kinetic chain continuity. The interventions include 1) an experimental intervention purported to engage muscles that naturally resist the collapsing effects of gravity, and 2) a control intervention designed to inhibit other muscle groups that are sometimes involved in maintaining bipedal alignment in a compensatory role. Study outcomes are measured before and after both interventions to quantify the acute effects of each. All participants complete both interventions in random order, crossing over after a one-week washout period. This research will provide insight into the acute effects of studied interventions, specifically those relating to maintenance of bipedal alignment with respect to gravitational collapsing tendencies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* 18 - 40 years of age

Exclusion Criteria:

* Recent (< 6 months) history of lower extremity injury
* Recent (< 6 months) history of other musculoskeletal or neurological disorder affecting balance
* Contraindications to participation in physical activity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Euclidean distance from the vector describing subject-specific, simulated gravitational collapse | Immediately before Intervention (Day 1)
  This outcome is a cumulative descriptor of segment angle distance from the pattern in which an individual's posture would collapse. The reference point for each individual is calculated using both pre and post-intervention data for a given day.
Euclidean distance from the vector describing subject-specific, simulated gravitational collapse | Immediately after Intervention (Day 1)
  This outcome is a cumulative descriptor of segment angle distance from the pattern in which an individual's posture would collapse. The reference point for each individual is calculated using both pre and post-intervention data for a given day.
Euclidean distance from the vector describing subject-specific, simulated gravitational collapse | Immediately before Intervention (Day 7)
  This outcome is a cumulative descriptor of segment angle distance from the pattern in which an individual's posture would collapse. The reference point for each individual is calculated using both pre and post-intervention data for a given day.
Euclidean distance from the vector describing subject-specific, simulated gravitational collapse | Immediately after Intervention (Day 7)
  This outcome is a cumulative descriptor of segment angle distance from the pattern in which an individual's posture would collapse. The reference point for each individual is calculated using both pre and post-intervention data for a given day.
Pooled intermuscular coherence | Immediately before Intervention (Day 1)
  Weighted average of frequency-domain correlations between muscle pairs belonging to anterior, posterior, and trunk muscle groups.
Pooled intermuscular coherence | Immediately after Intervention (Day 1)
  Weighted average of frequency-domain correlations between muscle pairs belonging to anterior, posterior, and trunk muscle groups.
Pooled intermuscular coherence | Immediately before Intervention (Day 7)
  Weighted average of frequency-domain correlations between muscle pairs belonging to anterior, posterior, and trunk muscle groups.
Pooled intermuscular coherence | Immediately after Intervention (Day 7)
  Weighted average of frequency-domain correlations between muscle pairs belonging to anterior, posterior, and trunk muscle groups.

SECONDARY OUTCOMES:
Top-down kinetic chain continuity | Immediately before Intervention (Day 1)
  The purpose of this outcome is to quantify the communication of motion from the upper body to the lower body. In a test involving placing hands-on-head and pulling the elbows back as far as possible, the response in the lower body is quantified by posterior rotation of the tibial segment.
Top-down kinetic chain continuity | Immediately after Intervention (Day 1)
  The purpose of this outcome is to quantify the communication of motion from the upper body to the lower body. In a test involving placing hands-on-head and pulling the elbows back as far as possible, the response in the lower body is quantified by posterior rotation of the tibial segment.
Top-down kinetic chain continuity | Immediately before Intervention (Day 7)
  The purpose of this outcome is to quantify the communication of motion from the upper body to the lower body. In a test involving placing hands-on-head and pulling the elbows back as far as possible, the response in the lower body is quantified by posterior rotation of the tibial segment.
Top-down kinetic chain continuity | Immediately after Intervention (Day 7)
  The purpose of this outcome is to quantify the communication of motion from the upper body to the lower body. In a test involving placing hands-on-head and pulling the elbows back as far as possible, the response in the lower body is quantified by posterior rotation of the tibial segment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Glass, PhD, Principal Investigator — Radford University
Locations (1):
- Radford University Carilion, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data for individual participants will be shared upon request with parties committing to institutional data sharing agreements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: On request and indefinitely.